CLINICAL TRIAL: NCT04724863
Title: Analysis of Respiration-induced Deformities of the Visceral and Renal Arteries Before and After Stenting for a Endovascular Aortic Repair Procedure Using a Fenestrated Prothesis
Brief Title: Analysis of Respiration-induced Deformities of the Visceral and Renal Arteries Before and After Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02417-50
Record Dates: First submitted 2020-03-10; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Complex Aortic Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol (Experimental): Each patient agreeing to participate in the study will be distributed in the protocol group and will receive an angioscan according to the protocol in pre-operative and at the usual post-operative check-up within 3 months after the operation. The usual procedure, foresees an angioscanner with injection of contrast product and the measurement of the images is performed during a deep breath. In order to obtain a complete respiratory cycle, the study procedure foresees in addition to the usual procedure, an image measurement during a deep exhalation.
  Interventions: Procedure: Angioscan

INTERVENTIONS:
Procedure: Angioscan — The study procedure foresees to take images during a deep breath as well as deep exhalation. This second measurement does not require the administration of an additional amount of contrast material. However, the exposure time to ionising radiation is doubled. The examination uses helical acquisition in fast mode. The duration of the helix is of the order of 2 seconds in the inspiration phase, then there is a delay of 5 seconds of machine time ("half-turn") and again 2 seconds of exposure in the expiration phase, i.e. 4 seconds of actual exposure to ionizing radiation, the time of image taking and 9 seconds the total time of the examination.

SUMMARY:
Fenestrated stents are used for the management of complex juxta-renal, para-renal or thoracoabdominal aneurysms in patients with high surgical risk and/or contraindicated for open surgery. These endovascular techniques have demonstrated their safety and efficacy, however, long-term follow-up CT scans remain essential for the detection of complications such as endo-leaks and restenosis/thrombosis of visceral and renal stents. The respiratory cycle might induce changes in the geometry and deformations of visceral and renal stents after complex aortic procedures. These could be detected by an adapted CT scan analysis by deep inhalation and deep exhalation acquisition carried out pre-operatively and post-operatively for monitoring of these same stents and screening for complications.

ELIGIBILITY:
Inclusion Criteria:

* no contre indication for coroscanner

Exclusion Criteria:

* pregnant woman
* allergy to iodinated contrast media
* vulnerable people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Geometry of the visceral and renal branches | 1 day
  An angioscanner will be performed with injection in inspiration and expiration (breathing cycle) before and after stent placement for a fenestrated aortic endografts.
  After reconstruction of a 3D volume of the aorta and extraction of the central lines of the different target arteries, the angle of the different visceral and renal branches will be measured during the respiratory cycle (inspiration; expiration) and compared before and after stenting.

SECONDARY OUTCOMES:
Endoleaks number | 3 months
stenosis number | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan HAULON, Pr, Study Director — Hopital Marie Lannelongue; Justine MOUGIN, Dr, Principal Investigator — Hopital Marie Lannelongue; Olaf MERCIER, Pr, Study Chair — Hopital Marie Lannelongue
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaoguo Y, Zhong C, Lei K, Yaowen X. Treatment of complex aortic aneurysms with fenestrated endografts and chimney stent repair: Systematic review and meta-analysis. Vascular. 2017 Feb;25(1):92-100. doi: 10.1177/1708538115627718. Epub 2016 Jul 10. PMID 26846442
- [Background] Eagleton MJ, Farivar B, Dias A. Large, single-center databases and the evolution of endovascular therapy for complex aortic aneurysms. Surgery. 2017 Nov;162(5):963-973. doi: 10.1016/j.surg.2017.03.018. Epub 2017 May 25. PMID 28552169
- [Background] Spear R, Sobocinski J, Hertault A, Delloye M, Azzauiu R, Fabre D, Haulon S. One Year Outcomes of 101 BeGraft Stent Grafts used as Bridging Stents in Fenestrated Endovascular Repairs. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):504-510. doi: 10.1016/j.ejvs.2018.01.023. Epub 2018 Mar 1. PMID 29501401
- [Background] Ullery BW, Suh GY, Lee JT, Liu B, Stineman R, Dalman RL, Cheng CP. Geometry and respiratory-induced deformation of abdominal branch vessels and stents after complex endovascular aneurysm repair. J Vasc Surg. 2015 Apr;61(4):875-84. doi: 10.1016/j.jvs.2014.11.075. Epub 2015 Jan 15. PMID 25601499